CLINICAL TRIAL: NCT06072937
Title: Clinical Evaluation of HeartPoint Global Intellistent for Pulmonary Flow Adjustment in Congenital Heart Disease and Dilated Cardiomyopathy
Brief Title: IntelliStent for Pulmonary Flow Adjustment in Congenital Heart Disease and Dilated Cardiomyopathy
Acronym: HEARTFUL-CHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HeartPoint Global (Industry)
Collaborators: Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPG-001-23
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Arterial Hypertension; Dilated Cardiomyopathy; Congenital Heart Disease
Keywords: pediatric cardiology; pulmonary arterial hypertension; dilated cardiomyopathy
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Cardiomyopathy, Dilated; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Single Arm Early Feasibility Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IntelliStent Arm (Experimental): Single Arm Safety and Effectiveness of the IntelliStent System
  Interventions: Device: IntelliStent

INTERVENTIONS:
Device: IntelliStent — Staged implantation of IntelliStent. The system comprises a nitinol self-expanding stent with a hollow element delivered over-the-wire into the main pulmonary artery or its left and right branches, using an 18 Fr transfemoral introducer sheath. The stent consists of two sections, one with a larger diameter and one with a smaller diameter, available in 6 sizes suitable for vessel sizes ranging from 20mm to 30 mm. Additional smaller sizes are currently under development.

SUMMARY:
IntelliStent is intended to achieve reduction of pulmonary hypertension, improvements in symptoms and quality of life in pediatric, adolescent and adult patients with congenital heart disease associated pulmonary arterial hypertension or left ventricular dilated cardiomyopathy.

DETAILED DESCRIPTION:
IntelliStent Implant System is a kit of stents for adjustable interventional reduction of blood flow through a novel and minimally invasive intervention to replace surgical Pulmonary Artery Banding (PAB).

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adolescent (12-17 years) or Adult (age >18 years)
2. Uncorrected CHD (ASD, VSD, PDA, AVSD) with left to right + systemic pulmonary artery pressure or mixed shunting regardless if pulmonary vascular resistance is modifiable or fixed
3. Diagnosed with WHO Group 1 PH Classification pulmonary hypertension associated with congenital heart disease, evidence by the following parameters measured at rest:

   1. Mean pulmonary artery pressure (mPAP) ≥ 50 mmHg
   2. Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP)

      ≤ 15 mmHg.
   3. Pulmonary vascular resistance > 3 Wood Units
4. Patients with left ventricular dilated cardiomyopathy with symptoms despite optimal medical therapy
5. Current WHO Functional Class III or IV.
6. Patients with the following anatomical dimensions (gated CT with angio or MRI with EKG) at target implantation site:

   1. MPA diameter @ systolic ≥ 15 mm and ≤ 24 mm and length @ systolic ≥ 28 mm, or
   2. Left and Right PA Branch diameter @ systolic ≥ 15 mm and ≤ 24 mm and length @ systolic ≥ 28 mm
7. Main pulmonary artery (MPA) or left/right PA Branch anatomy suitable for placement of the device as defined in the Instructions For Use (IFU) and as assessed by computed tomography (CT), fluoroscopy or echocardiography.
8. Each patient, or his or her guardian or legal representative, is willing to give informed consent, subject to national law.

Exclusion Criteria:

1. Right ventricular dysfunction
2. Severe AV valve regurgitation of the pulmonary ventricle
3. Complex CHD
4. Ongoing infection
5. Patients where definitive correction of the CHD is indicated and available as a possible treatment option
6. Patients with pressure gradient across the systemic outflow tract/subaortic region >40 mmHg @ rest
7. PAH-CHD patients with small defects that may be incidental findings
8. PAH after corrective cardiac surgery
9. Anatomical limitation to IntelliStent® (e.g. pulmonary artery size)
10. Known or suspected thrombosis of the femoral or iliac veins on the proposed site of venous cannulation
11. Vasculature lesions or characteristics that prevent percutaneous transluminal catheterization
12. Allergies or contraindications to prescribed procedural medications and contrast medium Anomalous pulmonary venous return (total or partial)
13. Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel
14. Mental incapacity, unwillingness or language barrier precluding adequate understanding of the trial procedure or cooperation with trial site personnel
15. Pregnant, lactating or planning pregnancy

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-04 (Estimated); Primary Completion 2025-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance (PVR) | 24 Weeks
  The primary efficacy endpoint is a binary variable. For patients with a baseline pulmonary vascular resistance (PVR) >1000 dynes·s·cm-5, success is defined by an absolute reduction in PVR of ≥300 dynes·s·cm-5 at 24 weeks. For patients with a baseline PVR ≤1000 dynes·s·cm-5, success is a 30% reduction in PVR at 24 weeks.

SECONDARY OUTCOMES:
Six Minute Walk Test Distance | 12 Weeks
  Change from baseline of six minute walk test distance (meters) at Week 12.
Change From Baseline to Week 12 in Borg Dyspnea Score | Baseline to 12 weeks
  The Borg Dyspnea score is a self-rating scale to evaluate the severity of dyspnea (from 0 "no shortness of breath at all" to 10 "very, very severe / maximal" shortness of breath).
NYHA Class change from Baseline at Week 12 | Baseline to 12 weeks
  New York Heart Association Class (NYHA) class: minimum I; maximum IV ( worse)
Change From Baseline to Week 12 in Ejection Fraction | Baseline to 12 Weeks
  Ejection Fraction (%) measured by transthoracic echocardiography
Change From Baseline to Week 12 in Left Ventricular Volumes | Baseline to 12 Weeks
  Left Ventricular Volumes measured by transthoracic echocardiography
Change From Baseline of the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to 12 Weeks
  KCCQ scores for quality of life are scaled from 0 to 100 and summarized in 25-point ranges: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent

CONTACTS AND LOCATIONS:
Overall Officials: Monica Tocchi, MD, PhD, Study Director — Meditrial USA Inc. Clinical Research Organization

IPD SHARING:
Plan to Share IPD: Yes
The dataset generated during and/or analysed during the study will be available upon request from the Clinical Research Organization, Meditrial USA Inc. m.tocchi@meditrial.net Datasets will only be made available through publication, unless disclosure is mandated by law
Time Frame: Intention to publish date 09/01/2024
Access Criteria: Available on request, Published as a supplement to the results publication.

REFERENCES:
- See also: Heartpoint Global — https://www.heartpointglobal.com/
- See also: Meditrial Clinical Research Organization — https://www.meditrial.net/